CLINICAL TRIAL: NCT03668834
Title: A Comparative Study Between Recipient Site Preparation Using Dermabrasion,Liquid Nitrogen Induced Blister and Dermarolling System in Autologous Non Cultured Epidermal Cell Suspension Procedure in Stable Vitiligo Patients.
Brief Title: Comparing Recipient Site Preparation Using Dermabrasion, Dermaroller and Liquid Nitrogen Induced Blister in Non Cultured Epidermal Cell Suspension in Stable Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Davinder Parsad, Dr.Davinder Parsad, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/TEC/2018/000424
Record Dates: First submitted 2018-06-27; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Dermabrasion

STUDY DESIGN:
Intervention Model Description: All 3 methods of recipient site preparation will be done in all 36 patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dermabrasion with NCES (Active Comparator): Intervention-Dermabrasion with autologous non cultured epidermal cell suspension Recipient site preparation using dermabrasion followed by autologous non cultured epidermal cell suspension technique of 1 stable vitiligo patch of each of the 36 patients.
  Interventions: Procedure: Dermabrasion with NCES
- Dermaroller with NCES (Active Comparator): Intervention-Dermaroller with autologous non cultured epidermal cell suspension Recipient site preparation using dermaroller system followed by autologous non cultured epidermal cell suspension technique of 1 stable vitiligo patch of each of the 36 patients.
  Interventions: Procedure: Dermaroller with NCES
- Liquid nitrogen induced blister with NCES (Active Comparator): Liquid nitrogen induced blister with autologous non cultured epidermal cell suspension Recipient site preparation using liquid nitrogen induced blister followed by autologous non cultured epidermal cell suspension technique of 1 stable vitiligo patch of each of the 36 patients.
  Interventions: Procedure: Liquid nitrogen induced blister with NCES

INTERVENTIONS:
Procedure: Dermabrasion with NCES — 1. The recipient site will be shaved, cleaned with betadine and surgical spirit and anaesthetized with mixture of 2% lignocaine and NS (1:1).
  2. Dermabrasion will be done using Manekshaw's dermabrader until tiny pinpoint bleeding spots are seen and extended 5mm beyond margins to prevent halo phenomenon.
  3. The denuded area will be washed with PBS and covered with a PBS moistened gauze piece.
  4. With 18 G needle attached to tuberculine syringe, few small drops of non cultured epidermal cell suspension will be placed over the denuded surface and spread evenly.
  5. Dressing is done in 4 layers in order-collagen(Neuskin F), bactigras, cutisoft(sterile gauze) and dynaplast (elastic plaster).
  Arms: Dermabrasion with NCES
Procedure: Dermaroller with NCES — 1. The recipient site will be shaved, cleaned with betadine and surgical spirit.
  2. Microneedling will be done with a device containing 540 microneedles in 8 rows, each 0.25 mm in length. Microneedling will be extended 5 mm beyond margins to prevent halo phenomenon.
  3. The roller will be passed repeatedly over the skin in a star-shaped way for about 10 minutes
  4. The noncultured epidermal cell suspension will be carefully transferred to a tuberculin syringe.
  5. NCES will be applied to the skin surface with a tuberculin syringe with an 18G needle and spread evenly after dermarolling treatment.
  6. Dressing is done in 4 layers in order-collagen(Neuskin F), bactigras, cutisoft(sterile gauze) and dynaplast (elastic plaster).
  Arms: Dermaroller with NCES
Procedure: Liquid nitrogen induced blister with NCES — 1. The recipient site will be shaved, cleaned with betadine and surgical spirit and anaesthetized with mixture of 2% lignocaine and NS (1:1).
  2. The site to be grafted is outlined with a surgical marking pen.
  3. To induce blisters on the achromic areas, freezing with liquid nitrogen spray was performed during 10 to 20 seconds inside round circles previously drawn on the skin.
  4. The patient is asked to visit 24 hours later.
  5. The blister fluid is aspirated and NCES taken in tuberculin syringe with 18 G needle is injected into it such that the blister roof is preserved.
  6. Dressing is done in 4 layers in order-collagen(Neuskin F), bactigras, cutisoft(sterile gauze) and dynaplast (elastic plaster).
  Arms: Liquid nitrogen induced blister with NCES

SUMMARY:
A COMPARATIVE STUDY BETWEEN RECEPIENT SITE PREPARATION USING DERMABRASION, LIQUID NITROGEN INDUCED BLISTER AND DERMAROLLING SYSTEM IN AUTOLOGOUS NON CULTURED EPIDERMAL CELL SUSPENSION PROCEDURE IN STABLE VITILIGO PATIENTS

DETAILED DESCRIPTION:
With a sample size of 36, 3 patches of a single stable vitiligo patient will be prepared using dermabrasion,dermaroller system and liquid nitrogen induced blister. The autologous non cultured epidermal cell suspension will be prepared using cold trypsinization from the skin graft taken from patient.After preparation of the recipient site,the suspension is applied and dressing is done.The patient is followed up for 3 months and extent of repigmentation,colour match,pattern of repigmentation,patient satisfaction score, vitiligo quality of life index before and after surgery and effect on acral vs non acral regions are studied for all the 3 methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of generalized vitiligo
* Patients with symmetrical lesions of size > 1.5cm x 1cm present on trunk or extremities including acral areas.
* Vitiligo lesions has been stable for 1 year.
* Disease not responding to medical treatment, or there are residual patches (after medical therapy) of vitiligo .
* Maximum size of vitiligo patches to be selected for surgery will not be >100cm2.

Exclusion Criteria:

* Age less than 18 years
* Pregnancy and lactation
* Patient with actively spreading vitiligo
* History of Koebnerisation
* History of hypertrophic scars or keloidal tendency
* Bleeding disorders
* Patients with unrealistic expectation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of extent of repigmentation in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non culured epidermal cell suspension. | 3 months from the surgery
  The extent of repigmentation is done by measurement of lesions in a tracer paper before and after surgery and comparison of pre operative and post operative images clicked in Canon Powershot SX620HS 20.2MP camera and grading is done as
  ≤25% Minimal repigmentation 26-50% Mild repigmentation 51-75% Moderate repigmentation 76-90% Marked repigmentation >90% Excellent repigmentation

SECONDARY OUTCOMES:
Comparison of colour match of repigmentation in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non culured epidermal cell suspension. | 3 months from the surgery
  Comaprison is done by matching the colur of repigmented skin with the colour of normal skin and grading it as 'somewhat lighter than', 'same as' or 'somewhat darker than' normal skin.
Comparison of pattern of repigmentation in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non cultured epidermal cell suspension. | 3 months from the surgery
  Comparison is done by using pre operarative and post operative images of the lesions clicked using Canon SX620HS 20.2 MP camera and classified as
  * Diffuse
  * Perifollicular
  * Migrating from the borders
Comparison of adverse events in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non cultured epidermal cell suspension. | 3 months from the surgery
  Recipient site adverse effects
  * infection
  * milia
  * scarring Donor site adverse effects
  * Infection
  * Milia
  * Scarring
  * Hypopigmentation
  * Hyperpigmentation
  * rejection
Comparison of repigmentation in acral vs non acral areas in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non cultured epidermal cell suspension. | 3 months from the surgery
  Repigmentation is compared between acral and non acral areas using pre operative and post operative images clicked by Canon SX620HS 20.2MP camera.
Patient satisfaction index | 3 months from the surgery
  Patients are asked to fill patient satisfaction index after surgery which is a questionaire with scores ranging from 0-30.
Vitiligo quality of life index. | 3 months from the surgery
  Comparison of vitiligo quality of life index before and after surgery in the vitiligo patches following dermabrasion, dermaroller system and liquid nitrogen induced blister followed by autologous non cultured epidermal cell suspension with scores ranging from 0-96.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided